CLINICAL TRIAL: NCT04268446
Title: Investigation of the Turkish Version, Validity and Reliability of Brief-BESTest Scale in Stroke Patients
Brief Title: Turkish Version of the Brief-BESTest Scale
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Kübra Uğurlu, Research Assistant, Kırıkkale University
Other Study IDs: turkishbriefBESTest
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Stroke Patients
Keywords: brief BESTest; stroke patients; Turkish version

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the validity and reliability of the Turkish version of the brief-BESTest (short BESTest) scale in stroke patients.

DETAILED DESCRIPTION:
Brief Balance Evaluation Systems Test (Brief-BESTest) is a short version of the Balance evaluation systems test (BESTest). Balance assessment systems test (BESTest) The balance assessment systems test developed by Horak consists of 6 sub-sections that evaluate the systems related to balance; 1) biomechanical limitations, 2) stability limit, 3) postural responses, 4) intuitive postural adjustments, 5) sensory orientation and 6) walking. It consists of 36 tests in total. Each question is rated between 0-3. The highest score that can be obtained is 108. Low test scores show that the balance is disturbed. BESTest has been found to be reliable among raters evaluating a cohort of individuals with and without various neurological diagnoses. In studies conducted, it was stated that BESTest is reliable when compared to other scales evaluating balance.

The necessary permissions have been obtained from the authors for Short BESTest, whose validity and reliability features will be tested, and the translation process to Turkish has been completed and the survey has been finalized. The basis for the use of special tools such as the scale is to prove the usability of the tool in the sample group to which it will be applied. The first step for this is the translation stage from the original language to the other language.

At the stage of translation into Turkish, two experts who knew a good level of English translated the questionnaire from English into Turkish. These translations have been translated back into Turkish by two native speakers of English and distant medical subjects. In addition, these translations were re-examined by the researchers and turned into a single form. This form was sent to five specialists in the field, checking the content and compliance with Turkish was evaluated. With the opinion of experts, the scale was finalized.

The study will include individuals over 40 years of age who have been diagnosed with an ischemic or hemorhagic stroke, who applied to the Kırıkkale University Faculty of Medicine Physical Therapy and Rehabilitation Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Being 40 years old or older,
* Diagnosis of stroke,
* No cooperation and communication problems
* To be able to walk 10 m independently with or without an auxiliary device

Exclusion Criteria:

* Another neurological or orthopedic problem other than stroke that will affect functionality and balance
* Individuals with advanced contraindications for cardiovascular disease and mobilization will not be included in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are able to walk 10 m independently with or without a device over 40 years old with a diagnosis of stroke.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Test | 15 minutes
  It is a 14-item scale that evaluates the tasks used in daily life activities.Standing up without support, standing without support, sitting without support, standing up, transfers, standing with feet, standing with legs while standing, reaching out while standing, picking up from the ground, looking back, 360 degree rotation, firm side standing on the stool, one foot standstill and standstill functions are evaluated.Each item is planned between 0-4; 0 is unable to fulfill the task, 4 is to fulfill the task successfully. The total score of the test is between 0-56.0-20 points: wheelchair dependent, 21-40: assisted walking, 41-56: means independent ambulation.
Functional Reach Test | 5 minutes
  Subjects will asked to stand comfortably, to make a fist, and to raise their arm until it was parallel to the yardstick (position 1). The placement of the end of the third metacarpal along the yardstick will recorded. Subjects will then asked to reach as far forward as they could without losing their balance (position 2), and the position of the end of the third metacarpal along the yardstick will again recorded. No attempt will make to control the subject's method of reach, but if he will touch the wall or took a step during the maneuver, that trial will consider invalid and repeated.
Time Up and Go Test | 5 minutes
  This test is applied to assess the risk of falling and mobility.This test starts with the individual leaving the chair without receiving arm support by giving the go command while sitting in a chair.The distance of 3 meters is asked to return and sit again in the chair.The elapsed time is recorded in seconds.
10 Meter Walk Tests | 3 minutes
  Walking speed are measure by timing subjects over 10 meters with a stopwatch. To avoid the effects of acceleration and deceleration, measurements take over the middle 10 meters of a 14-meter walkway. It is repeated 2 times.
Falls Efficacy Scale | 5 minutes
  FES is a 10-item scale and these items are; To enter and get out of bed, to sit and stand on the chair, to take a bath or shower, to dress and undress, to lie on the shelves, to walk in the house, to answer the door or phone, to prepare food without lifting heavy objects and to do simple shopping. Individuals score between 0 (not safe) and 10 (very safe) for each question, and when all scores are summed, a total score between 0 and 100 is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Saniye Aydoğan Arslan, Study Director — Kırıkkale University; Kübra Uğurlu, Principal Investigator — Kırıkkale University; Cevher Demirci, Principal Investigator — Balikesir University; Zekiye İpek Katırcı Kırmacı, Principal Investigator — Sanko University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padgett PK, Jacobs JV, Kasser SL. Is the BESTest at its best? A suggested brief version based on interrater reliability, validity, internal consistency, and theoretical construct. Phys Ther. 2012 Sep;92(9):1197-207. doi: 10.2522/ptj.20120056. Epub 2012 Jun 7. PMID 22677295
- [Background] Smith PS, Hembree JA, Thompson ME. Berg Balance Scale and Functional Reach: determining the best clinical tool for individuals post acute stroke. Clin Rehabil. 2004 Nov;18(7):811-8. doi: 10.1191/0269215504cr817oa. PMID 15573838
- [Background] Schmidt S, Bullinger M. Current issues in cross-cultural quality of life instrument development. Arch Phys Med Rehabil. 2003 Apr;84(4 Suppl 2):S29-34. doi: 10.1053/apmr.2003.50244. PMID 12692769
- [Background] Chinsongkram B, Chaikeeree N, Saengsirisuwan V, Viriyatharakij N, Horak FB, Boonsinsukh R. Reliability and validity of the Balance Evaluation Systems Test (BESTest) in people with subacute stroke. Phys Ther. 2014 Nov;94(11):1632-43. doi: 10.2522/ptj.20130558. Epub 2014 Jun 12. PMID 24925073
- [Background] Bergstrom M, Lenholm E, Franzen E. Translation and validation of the Swedish version of the mini-BESTest in subjects with Parkinson's disease or stroke: a pilot study. Physiother Theory Pract. 2012 Oct;28(7):509-14. doi: 10.3109/09593985.2011.653707. Epub 2012 Jan 30. PMID 22288658
- [Background] O'Hoski S, Sibley KM, Brooks D, Beauchamp MK. Construct validity of the BESTest, mini-BESTest and briefBESTest in adults aged 50 years and older. Gait Posture. 2015 Sep;42(3):301-5. doi: 10.1016/j.gaitpost.2015.06.006. Epub 2015 Jun 25. PMID 26183191
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] Horak FB, Wrisley DM, Frank J. The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther. 2009 May;89(5):484-98. doi: 10.2522/ptj.20080071. Epub 2009 Mar 27. PMID 19329772